CLINICAL TRIAL: NCT07199218
Title: A Phase 2, Placebo-Controlled, Randomized, Double-Blind Study to Assess the Safety, Tolerability and Efficacy of Terpenes-enriched Cannabis Oil T1/C28, Administered to Pediatric Subjects With Autism Spectrum Disorder (ASD)
Brief Title: Placebo-Controlled Study of Terpenes-Enriched Cannabis Oil T1/C28 for Children With Autism
Acronym: TECA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bazelet Nehushtan LtD. (Industry)
Responsible Party: Principal Investigator, Adi Aran, Director, Neuropediatric unit, SZMC, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0336-24-SZMC; MOH_2025-04-21_014042 (Registry Identifier: Clinical Trials.gov.il)
Record Dates: First submitted 2025-09-11; First posted 2025-09-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; ASD; cannabidiol; terpenes; THC
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terpenes-Enriched CBD-Predominant Oil (Experimental): Oral cannabidiol (CBD), tetrahydrocannabinol (THC; 1/28 of the CBD dose), and terpenes, administered for 8 weeks as an add-on to existing treatments. After the first 8 weeks, participants will continue with the same treatment for an additional 8 weeks.
  Interventions: Drug: Terpenes-Enriched CBD-Predominant Oil
- Placebo (Placebo Comparator): Oral olive oil with flavoring to mimic the texture and taste of the study drug, given for 8 weeks. After the first 8 weeks, participants will switch to terpenes-enriched CBD oil without THC for another 8 weeks.
  Interventions: Drug: Placebo; Drug: Terpenes-Enriched CBD Oil (THC-Free)

INTERVENTIONS:
Drug: Terpenes-Enriched CBD-Predominant Oil — Oral cannabidiol (CBD; 7.2 mg/kg/day), tetrahydrocannabinol (THC; 0.257 mg/kg/day, equivalent to 1:28 of the CBD dose), and terpenes (0.5 mg/kg/day), administered in two daily doses. The formulation is an olive oil-based solution (CBD/THC: 280/10 mg per g) produced by Bazelet Group, Israel.
  Arms: Terpenes-Enriched CBD-Predominant Oil
Drug: Placebo — Oral olive oil with added flavors to mimic the appearance, texture, and taste of the study drug, administered in two daily doses.
  Arms: Placebo
Drug: Terpenes-Enriched CBD Oil (THC-Free) — Oral cannabidiol (CBD; 7.2 mg/kg/day) and terpenes (0.5 mg/kg/day), administered in two daily doses. The formulation is an olive oil-based solution (CBD- 280 mg per g) produced by Bazelet Group, Israel.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine whether cannabidiol (CBD, 28%) combined with terpenes and a small amount of THC (1%) can help reduce symptoms of autism, and to evaluate the safety of this treatment.

The main questions are:

1. Does this treatment improve behavioral challenges in children with autism?
2. Does this treatment improve social difficulties in children with autism?

What will happen in the study:

1. Participants take either the study treatment or a placebo (a look-alike substance with no active drug) every day for 2 months.
2. After 2 months, all participants receive the study treatment or a similar treatment without THC for another 2 months.
3. Participants come to the clinic once every 2 months for checkups and tests.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a condition that affects communication, social interaction, and behavior. Current medications do not treat the core symptoms of autism, and the drugs sometimes prescribed (such as antipsychotics for irritability) can cause significant side effects.

Cannabidiol (CBD) is a natural, non-psychoactive compound from the cannabis plant that may reduce brain overactivity and inflammation. Tetrahydrocannabinol (THC), the psychoactive component of cannabis, acts on the endocannabinoid system, which is thought to function differently in people with autism. Research suggests that CBD combined with very small amounts of THC may improve behavior and social functioning. Other plant compounds called terpenes may enhance the effects of CBD and THC, even at low doses.

This study tests whether a CBD oil enriched with terpenes and a very small amount of THC is safe and effective for children with autism. Seventy-eight children, ages 4-13, will participate. Half will receive the study oil and half will receive a placebo (an inactive oil that looks the same) for 8 weeks. Afterward, all participants will receive an active treatment for another 8 weeks.

The study evaluates whether the treatment improves behavior, social skills, and quality of life. Safety is monitored through regular clinic visits, questionnaires, physical exams, and blood tests.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4 to 12 years (after the 4th birthday and before the 13th).
2. Diagnosis of autism spectrum disorder (ASD) according to DSM-5, confirmed by Childhood Autism Rating Scale-Second Edition (CARS-2).
3. Moderate or greater ASD-associated symptoms, defined as a rating of ≥4 ("moderate" or higher) on the Overall Function Clinical Global Impression-Severity (CGI-S).
4. Aberrant Behavior Checklist-Irritability subscale (ABC-I) score ≥18.
5. Social Responsiveness Scale-Second Edition (SRS-2) total T score ≥66.

Exclusion Criteria:

1. Body weight <12.5 kg or ≥57.5 kg.
2. Current or past diagnosis of heart failure, drug addiction, schizophrenia, psychosis, bipolar disorder, post-traumatic stress disorder (PTSD), or major depressive disorder (MDD), or diagnosis of schizophrenia in a first-degree relative.
3. Seizure or change in antiepileptic medications within 4 months prior to randomization.
4. Clinically significant abnormalities on physical examination or laboratory testing, including impairment in cardiac, hepatic, or renal function.
5. Change in pharmacological or behavioral treatment, or change in home or school environment (other than school holidays), within 4 weeks prior to randomization or planned during the study.
6. Cannabinoid treatment within 4 weeks prior to randomization.
7. Predicted poor compliance with study procedures (e.g., blood tests).
8. Concurrent use of opiates or alcohol.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Aberrant Behavior Checklist-Community (ABC-C): Irritability Subscale raw score (ABC-I) | Baseline to Week 8
  The ABC-C is a caregiver-completed questionnaire with 58 items, divided into five subscales. The ABC-I (Irritability) subscale includes 15 items that assess emotional and behavioral symptoms of ASD, such as aggression toward others, deliberate self-injury, temper tantrums, depressed mood, and rapidly shifting moods. Scores on this subscale range from 0 to 45, with higher scores indicating greater severity. Change from baseline to Week 8 is reported, with lower scores reflecting clinical improvement.

SECONDARY OUTCOMES:
Change From Baseline in Vineland™-III Adaptive Behavior Scales (VABS3) Socialization Domain Standard Score | Baseline to Week 8
  The VABS-3 Socialization domain measures interpersonal relationships, play and leisure, and coping skills, reflecting the individual's ability to engage in age-appropriate social interactions. Higher scores indicate better adaptive social functioning.
Change From Baseline in Social Responsiveness Scale-2nd edition (SRS-II) total raw score | Baseline, Weeks 8 and 17
  The SRS-2 measures the severity of social impairment associated with autism spectrum disorder. It includes five subscales: Social Awareness (8 items), Social Communication (22 items), Social Cognition (12 items), Social Motivation (11 items), and Restricted Interests and Repetitive Behavior (12 items). Two summary scores are derived: the Total Score (sum of all five subscales) and the Social Communication and Interaction (SCI) score, which combines the four social subscales excluding Restricted Interests and Repetitive Behavior. The SCI and RRB correspond to the two DSM-5 symptom domains of autism spectrum disorder. Raw scores range from 65 to 260; higher scores indicate greater severity of social impairment.
Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) | Baseline to Week 17
  Participants experiencing at least one adverse event that newly appeared or worsened after treatment initiation. Adverse events are graded as mild, moderate, or severe; hospitalizations are documented as serious adverse events; causality is categorized from not related to definitely related.
Number of Participants With Clinically Significant Abnormal Laboratory Values | Week 8
  Number of participants with clinically significant abnormal values in complete blood count (CBC), liver transaminases, or total bilirubin levels, as determined by the investigator.
Change From Baseline in Body Mass Index (BMI) | Baseline, Weeks 8 and 17
  Difference between baseline and week 8 body mass index (kg/m²)
Clinical Global Impressions-Improvement (CGI-I) Score | Weeks 8 and 17
  CGI-I is a clinician rating of overall change from baseline; scores range from 1 to 7, with higher scores indicating worse outcome; anchors: 1 very much improved; 2 much improved; 3 minimally improved; 4 no change; 5 minimally worse; 6 much worse; 7 very much worse.
Caregiver Global Impression of Change (CGIC or CaGC) | Weeks 8 and 17
  CGIC (CaGC) is a caregiver rating of overall change from baseline; scores range from 1 to 7, with higher scores indicating worse outcome; anchors: 1 very much improved; 2 much improved; 3 minimally improved; 4 no change; 5 minimally worse; 6 much worse; 7 very much worse.

OTHER OUTCOMES:
Change From Baseline in Aberrant Behavior Checklist-Community (ABC-C): Irritability Subscale raw score (ABC-I) | Baseline, Week 17
  Appears above
Change From Baseline in Vineland™ Adaptive Behavior Scales (VABS-3) Communication Domain Score | Baseline to Week 8
  The VABS-3 Communication domain measures receptive, expressive, and written language skills. Higher Communication scores indicate better adaptive functioning
Change From Baseline in Vineland™ Adaptive Behavior Scales (VABS-3) Maladaptive Behavior Domain Score | Baseline to Week 8
  The VABS-3 Maladaptive Behavior domain measures internalizing, externalizing, and other maladaptive behaviors. Higher Maladaptive Behavior scores indicate greater difficulties.
Change From Baseline in Emotion Dysregulation Inventory (EDI) | Baseline, Weeks 8 and 17
  The EDI measures the intensity and reactivity of emotional responses, reflecting difficulties with emotion regulation; scores range from 0 to 120, with higher scores indicating greater emotion dysregulation.
Change From Baseline in Multidimensional Assessment of Disruptive Behavior (MAP-DB) | Baseline, Weeks 8 and 17
  The MAP-DB assesses temper loss, aggression, noncompliance, and impulsivity, capturing the frequency and severity of disruptive behaviors. Higher scores indicate greater disruptive behavior.
Change From Baseline in Autism Impact Measure (AIM) | Baseline. Weeks 8 and 17
  The AIM assesses the frequency and impact of core autism symptoms in daily life. Higher scores indicate greater symptom frequency and impact.
Change From Baseline in Quality of Life in Autism Questionnaire (QOLA) total score | Baseline, Weeks 8 and 17
  The QOLA Parent version includes Part A, parents' overall perception of their quality of life, and Part B, the impact of ASD symptoms on parents' quality of life; higher scores indicate better quality of life. Total scores: Part A ranges from 28 to 140, with higher scores reflecting better perceived parental quality of life; Part B ranges from 20 to 100, with higher scores indicating that the child's autism-related difficulties are perceived as less problematic for the parent.
Change From Baseline in Children's Sleep Habits Questionnaire (CSHQ) | Baseline, Weeks 8 and 17
  he CSHQ assesses common sleep problems in children across multiple domains; scores range from 33 to 99, with higher scores indicating a greater likelihood of sleep problems.
Change From Baseline in Gastrointestinal Signs and Symptoms Inventory | Baseline, Weeks 8 and 17
  This inventory assesses the presence and severity of gastrointestinal problems such as constipation, diarrhea, abdominal pain, and bloating. Higher scores indicate greater gastrointestinal symptom burden.
Change From Baseline in Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, Weeks 8 and 17
  The BRIEF evaluates executive functioning in daily life, including working memory, inhibitory control, and cognitive flexibility. Higher scores indicate greater executive dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, N/A = Not Applicable, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the results of this trial will be made available to qualified researchers after study completion and publication of the primary results. Data will include baseline characteristics, outcome measures, and safety data.
  Supporting Information:
  Data will be shared beginning 12 months after publication and available for up to 5 years. Access will be granted upon submission of a methodologically sound proposal and approval by the principal investigator and institutional ethics committee. A data use agreement will be required to ensure protection of participant confidentiality. Supporting documents such as the study protocol and statistical analysis plan will also be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study protocol, statistical analysis plan (SAP), and informed consent form (ICF) are available prior to enrollment of the first participant. De-identified individual participant data and the clinical study report (CSR) are available beginning 12 months after publication of the primary results and remain available for up to 5 years.
Access Criteria: The study protocol, statistical analysis plan (SAP), and informed consent form (ICF) are available to the public prior to enrollment of the first participant. De-identified individual participant data (baseline characteristics, outcome measures, and safety data) and the clinical study report (CSR) are available to qualified researchers beginning 12 months after publication of the primary results. Access requires submission of a methodologically sound proposal, approval by the principal investigator and ethics committee, and execution of a data use agreement.

REFERENCES:
- Available data/document: Study Protocol — https://osf.io/f69ds/files/osfstorage — Study protocol, statistical analysis plan, and parental informed consent form are available in the OSF repository: https://osf.io/f69ds/files/osfstorage (Updated September 2025)
- Available data/document: Statistical Analysis Plan — https://osf.io/f69ds/files/osf — Study protocol, statistical analysis plan, and parental informed consent form are available in the OSF repository: https://osf.io/f69ds/files/osfstorage (Updated September 2025)
- Available data/document: Informed Consent Form — https://osf.io/f69ds/files/osf

DOCUMENTS (3):
  • Study Protocol (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT07199218/Prot_003.pdf
  • Statistical Analysis Plan (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT07199218/SAP_004.pdf
  • Informed Consent Form (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT07199218/ICF_002.pdf